Official Title: Clinical Results of Minimally Invasive Plate Osteosynthesis Versus Conventional Approach in Volar Locking Plate for Close Fractures of Distal End Radius Under WALANT

Study protocol

**Material and Methods** 

1. Patient

The Consolidated Standards of Reporting Trials (CONSORT) statement guidelines were followed in this single-

center, prospective, parallel group, assessor-blinded, randomized controlled trial. All procedures were approved by

the institutional review board of Police general hospital.

Patients who were diagnosed isolated closed fracture of distal end radius at Police General Hospital, Bangkok,

Thailand between October 2021 and February 2023 were divided into the conventional group and the MIPO group

at recruitment, using a computer-generated randomization program from www.randomizer.org. Patients were

informed about the treatment options during a pre-interviewing session, and all eligible patients gave their written

informed consent before the randomization and initialization of the allocated treatment. When patients arrived in

the operating room, randomization took place using sealed envelopes containing assigned numbers. These

envelopes were in the operating room and remained unopened until the patient's arrival. Neither the patient nor

the attending physicians were informed about the randomization process. The orthopedic surgeon who assessed

patient eligibility was not involved in randomization, thereby securing allocation concealment.

Inclusion criteria:

-We included those diagnosed with isolated closed fractures of the distal end radius requiring surgery,

-aged 18 years and older.

The Exclusion criteria were:

(1) Patients with bone fractures lasting more than 21 days

(2) open fractures

1

[Unique Protocol ID: Dh3108103/64] (October 5, 2021)

Official Title: Clinical Results of Minimally Invasive Plate Osteosynthesis Versus Conventional Approach in Volar Locking Plate for Close Fractures of Distal End Radius Under WALANT

(3) articular multifragmentary comminuted fractures of the distal radius categorized as AO/OTA 2R3C3

(4) not suitable to undergo volar approach surgery

(5) individuals with combined carpal fractures or dislocation

(6) ulna fractures

(7) associated injuries

(8) a history of previous wrist surgery

(9) diabetes mellitus

(10) chronic wrist inflammation

(11) wrist bone deformities

(12) the use of anticoagulation drugs

(13) uncooperative behavior

(14) those refusing to participate in the research

### 2. Methods

According to the WALANT solution in our institute (Jaroenporn et al., 2022), the steps for preparing the solution are as follows (Figure 2A). Firstly, 40 ml of 1% Lidocaine with adrenaline (1:100,000) and 10 ml of 0.5% Marcaine are added to the solution. Marcaine, a long-acting local anesthetic, helps prolong the duration of pain relief.

Additionally, 40 ml of Normal Saline Solution (NSS) is included; NSS acts as a diluent and ensures the appropriate volume of the anesthetic solution. Finally, 4 ml of 7.5% NaHCO3 (sodium bicarbonate) is added to balance the acid-base pH. By following these steps, a total solution volume of 94 ml is prepared.

Locking Plate for Close Fractures of Distal End Radius Under WALANT

All patients underwent volar locking plate fixation under WALANT. First, the periosteum of the radius is infiltrated at three different points: proximal, middle, and distal (radial styloid), with each point receiving 10 ml of anesthesia. This ensures that the circumferential periosteum of the radius bone is adequately anesthetized. Next, a subcutaneous infiltration along the volar skin incision of 10 ml is injected (Figure 2B). After a 30-minute period of allowing the anesthesia to take effect

Operative Procedure for MIPO:

The patient, under WALANT, was in the supine position on the surgical table. A minimal 2 cm skin incision was made on the volar side of the wrist, proximal to the wrist crease 2 cm. The Trans flexor carpi radialis approach (Trans FCR) was performed, and the surgical plane was dissected using curved scissors to increase exposure. To mobilize and protect the flexor carpi radialis (FCR) and flexor pollicis longus (FPL) ulnarly, a self-retractor was employed. Care was taken to avoid damaging the radial artery on the radial side and the palmar cutaneous branch of the median nerve on the ulnar side. The distal aspect of the pronator quadratus muscle was elevated using a periosteal elevator. A partial transverse cut was made in the pronator quadratus muscle at the distal end to approach the fracture site. Closed reduction and temporary fixation with K-wires were used to assist in the reduction. The alignment was checked under fluoroscopy. The DePuy Synthes VA-LCP Two-Column Distal Radius Plates 2.4, volar, narrow, with 6 head holes and a width of 19.5 mm (Synthes USA Products, LLC), were utilized in the procedure. These plates were chosen for their minimal width, allowing easy insertion through a small incision. One cortical screw was inserted into an elongate hole, followed by the insertion of 4 distal locking screws. An additional proximal vertical mini incision of 1 cm was made for fixation with 2 proximal locking screws. No drain was inserted, and cast immobilization was not required.

Post-operation:

Adhering to post-operative protocols, no drain was inserted, and cast immobilization was unnecessary. Immediate encouragement of active finger and wrist motion was provided after the operation. Both groups were administered pain medication for 7 days, including Tramadol (50 mg), 1 tablet three times daily; Naproxen (250 mg), 1 tablet twice daily; and Tolperisone (50 mg), 1 tablet three times daily. In cases where the patient's Visual Analog Scale (VAS) pain score exceeded 5, a 3 mg IV dose of morphine was administered as needed by the patient.

As part of their early post-operative rehabilitation, patients were instructed in the six-pack exercise and wrist range of motion (ROM) exercises.

#### 3. Evaluation

The data collector, an orthopedic resident unaware of the surgical technique used, obtained information. Neither the collector nor the patients observed the surgical incision.

The primary outcome was measured using the pain visual analogue scale (VAS). Regarding the pain VAS, a score of 0 indicated no pain, and a score of 10 indicated the worst imaginable pain. The pain VAS score was recorded in the morning first 7 day then in the 2nd, 6th, 10th, 14th, and 24th weeks after surgery.

Patients attended outpatient department (OPD) follow-up appointments in the 2nd, 6th, 10th, 14th, and 24th weeks after surgery. The Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH) score indicated a functional outcome. The patient's satisfaction, along with the cosmetic score (rating the scar's appearance on a scale of 0 to 5, with 5 being excellent),. Hand grip strength was measured as a percentage of the strength in the other hand using a baseline hydraulic hand dynamometer with a JAMAR device (lbs force) from Sammons Preston, Inc., Bolingbrook, IL 60440-4989, in a 90 degree raised and extended arm position. The patient squeezed the dynamometer three times, and the highest score was recorded. Pinch strength was assessed by raising the patient's arm in front of them and bending it at a 90-degree angle, testing with a JAMAR Hydraulic Pinch Gauge. Three pinches on the device provided the highest score.

### **4 Statistical Analysis**

IBM SPSS Statistics 27.0 was utilized for statistical analysis. Results were expressed as the mean ± standard deviation. Statistically significant differences were determined based on P < 0.05 and the 95% confidence interval (CI). The Fisher's exact test was used to evaluate baseline characteristics including sex, fracture side, cause, AO/OTA type. The paired t-test was used to evaluate the age, incision length, VAS pain score, Quick DASH, functional outcomes (grip, pinch strength, range of motion), operative time, Aesthetics, Satisfaction and radiographic parameters. All subjects were analyzed and none of the subjects were lost to follow-up.

# **CONSORT diagram**



## **Method**



- · Police General Hospital, Thailand
- October 2021 February 2023

# **Data collection process**

## 1) Pain Visual Analog Score

Pain Rating Scale - Wong-Baker FACES™ & Visual Analogue Scale (VAS)

### Wong-Baker FACES™ Pain Rating Scale



Source: Pain assessment in children undergoing venipuncture: The Wong-Baker faces scale versus skin conductance fluctuations - Scientific Figure on ResearchGate. Available from: https://www.researchgate.net/figure/Wong-Baker-Faces-TM-Pain-Rating-Scale-Reproduced-with-Permission-of-the-Wong-Baker-Faces\_fig1\_236604762 [accessed 12 Feb, 2020]

[6] Tries work by Department of Pharmacology and Pharmacy, HKU is licensed under a <u>Creative Commons Attribution-NonCommercial 3.0 Hong Kong License</u>. Last updated Feb 2020.

| Postoperative day | date | Pain VAS |
|-------------------|------|----------|
| 0 | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| 5 | | |
| 6 | | |
| 7 | | |

## 2) QuickDASH form

| | Qı | iick <b>DAS</b> | H | | | |
|---|---|---|---|---|---|---|
| Plea | se rate your ability to do the following activities in | the last week b | y circling the i | number below th | ne appropriat | e response. |
| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | UNABLE |
| 1. | Open a tight or new jar. | 1 | 2 | 3 | 4 | 5 |
| 2. | Do heavy household chores (e.g., wash walls, floors). | 1 | 2 | 3 | 4 | 5 |
| 3. | Carry a shopping bag or briefcase. | 1 | 2 | 3 | 4 | 5 |
| 4. | Wash your back. | 1 | 2 | 3 | 4 | 5 |
| 5. | Use a knife to cut food. | 1 | 2 | 3 | 4 | 5 |
| 6. | Recreational activities in which you take some force or impact through your arm, shoulder or hand (e.g., golf, hammering, tennis, etc.). | 1 | 2 | 3 | 4 | 5 |
| | | NOT AT ALL | SLIGHTLY | MODERATELY | QUITE<br>A BIT | EXTREMELY |
| 7. | During the past week, to what extent has your arm, shoulder or hand problem interfered with your normal social activities with family, friends, neighbours or groups? | 1 | 2 | 3 | 4 | 5 |
| | | NOT LIMITED<br>AT ALL | SLIGHTLY<br>LIMITED | MODERATELY<br>LIMITED | VERY<br>LIMITED | UNABLE |
| 8. | During the past week, were you limited in your work or other regular daily activities as a result of your arm, shoulder or hand problem? | 1 | 2 | 3 | 4 | 5 |
| | ise rate the severity of the following symptoms<br>ne last week. (circle number) | NONE | MILD | MODERATE | SEVERE | EXTREME |
| 9. | Arm, shoulder or hand pain. | 1 | 2 | 3 | 4 | 5 |
| 10. | Tingling (pins and needles) in your arm, shoulder or hand. | 1 | 2 | 3 | 4 | 5 |
| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | SO MUCH<br>DIFFICULTY<br>THAT I<br>CAN'T SLEEP |
| 11. | During the past week, how much difficulty have you had sleeping because of the pain in your arm, | 1 | 2 | 3 | 4 | 5 |

A QuickDASH score may not be calculated if there is greater than 1 missing item.

## 3) Table data collection

| | MIPO | Conventional | p-value |
|-----------------------|------|--------------|---------|
| Mean age, (SD); range | | | |
| Sex | | | |
| female | | | |
| male | | | |
| fracture side | | | |
| Dominant Hand | | | |
| Non-dominant Hand | | | |
| Cause | | | |
| fall | | | |
| road traffic accident | | | |
| sports | | | |
| AO/OTA 23 | | | |
| A2 | | | |
| A3 | | | |
| В3 | | | |
| C1 | | | |
| C2 | | | |

| | wk 2 | wk 6 | wk 10 | wk 14 | wk 24 |
|-----------------------|-------|-------|-------|-------|-------|
| (lbs) | F/U 1 | F/U 2 | F/U 3 | F/U 4 | F/U 5 |
| Grip strength Fx | | | | | |
| Grip strength normal | | | | | |
| Pinch strength Fx | | | | | |
| Pinch strength normal | | | | | |
| ROM Fx | | | | | |
| Flexion | | | | | |
| Extension | | | | | |
| Supination | | | | | |
| Pronation | | | | | |
| Radial deviation | | | | | |
| Ulnar deviation | | | | | |
| Pain (0-10) | | | | | |
| QuickDASH | | | | | |
| Wound size (mm) | | | | | |
| Cosmetic score | | | | | |
| Satisfy score | | | | | |

| | MIPO | Conventional | P-value |
|--------------------------|------|--------------|---------|
| Pain score | | | |
| Q-DASH score | | | |
| Grip strength | | | |
| Subjective cosmetic | | | |
| Satisfaction | | | |
| Volar tile | MIPO | Conventional | P-value |
| Initial | | | |
| Immediate post operation | | | |
| Final | | | |
| Radial inclination | MIPO | Conventional | P-value |
| Initial | | | |
| Immediate post operation | | | |
| Final | | | |
| Ulnar variance | MIPO | Conventional | P-value |
| Initial | | | |
| Immediate post operation | | | |
| Final | | | |

| patient | Pain (0-10) | | | | | | | | | | | | | Pain (0-10) mo | | | | | | | C | -DASH | (0-100 | 0) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (no #) | Pre | D1 | D2 | D3 | D4 | D5 | D6 | D7 | wk2 | wk6 | wk10 | wk14 | wk24 | (mg) | Pre | wk2 | wk6 | wk10 | wk14 | wk24 | | | | |

| patient | X-ray | | | | | | | | | | | Hand onin | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | RI | | UV | | | VT | | | Cos | Cos Sat | | Hand grip | | | |
| (no #) | Pre | Post | F/U | Pre | Post | F/U | Pre | Post | F/U | | | wk2 | wk6 | wk10 | wk14 | wk24 |